CLINICAL TRIAL: NCT07111559
Title: A Multicenter Randomized Controlled Trial Comparing Tissue Plasminogen Activator With Dual Antiplatelet Therapy for Patients With Hyperacute Single Perforating Artery Infarction
Brief Title: Lacunar Stroke hyperAcute Clinical Utilization of Novel Approach Regimens: Rt-PA vs. DAPT Randomised Clinical Trial
Acronym: LACUNAR-tPA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nippon Medical School (Other)
Collaborators: Japan Research Foundation for Clinical Pharmacology (Unknown); Takeda Science Foundation - Medical Research Grant (Unknown)
Responsible Party: Principal Investigator, Yuki Sakamoto, Associate Professor, Nippon Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMS-M-2024-210
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Lacunar Stroke; Stroke; Ischemic Stroke
Keywords: rt-PA; tissue-plasminogen activator; DAPT; dual antiplatelet therapy
MeSH Terms: conditions — Stroke, Lacunar; Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rt-PA (Active Comparator)
  Interventions: Drug: rt-PA
- DAPT (Experimental)
  Interventions: Drug: DAPT

INTERVENTIONS:
Drug: rt-PA — Recombinant tissue-plasminogen activator treatment. Low-dose (0.6mg/kg) alteplase will be given because this dosage is the only dosage approved in Japan.
  Arms: rt-PA
Drug: DAPT — Dual antiplatelet therapy with aspirin 200mg and clopidogrel 300mg.
  Arms: DAPT

SUMMARY:
The goal of this clinical trial is to learn if a combination of antiplatelet drugs works better than intravenous tissue plasminogen activator to treat small ischemic stroke (lacunar stroke). The main questions it aims to answer are:

Is a combination of antiplatelet drugs non-inferior to the current standard tissue plasminogen activator treatment? Does a combination of antiplatelet drugs reduce the bleeding complications than tissue plasminogen activator?

Researchers will compare a combination of antiplatelet drugs to tissue plasminogen activator to see if a combination of antiplatelet drugs works to treat small ischemic stroke (lacunar stroke).

Participants will:

Take a combination of antiplatelet drugs or be given intravenous tissue plasminogen activator Check the neurological status 3 months after stroke, in-person, by phone, or by mail.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Acute ischemic stroke within 4.5 hours from onset. If onset time is unknown because of impaired consciousness or aphasia, use the "last known well" time.
* A single perforating-artery infarct on brain MRI:

located in the corona radiata, putamen, internal capsule, thalamus, or pons; solitary, mainly round or oval, with a maximum diameter ≤ 20 mm; lesions only in the centrum semiovale are not allowed, but extension from the above sites into the centrum semiovale is allowed.

* No disability in daily life before the stroke (modified Rankin Scale ≤ 1).
* National Institutes of Health Stroke Scale (NIHSS) score ≤ 5.
* Written informed consent obtained.

Exclusion Criteria:

* Antithrombotic therapy considered inappropriate because of active bleeding, low platelet count, or similar conditions.
* Any contraindication to intravenous rt-PA, without blood pressures.
* ≥ 50 % stenosis or occlusion of the artery responsible for the stroke * (see note below).
* Diseases that require anticoagulation (e.g., atrial fibrillation, deep-vein thrombosis) *
* Inability to take medicine orally.
* Any other reason judged by the principal investigator or co-investigators to make participation inappropriate.

Note: This study targets hyper-acute stroke within 4.5 hours. To avoid treatment delay, items marked with * must be judged using the similar examinations that each site normally performs before rt-PA administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Excellent outcome | 3 months after stroke
  Modified Rankin scale score of 0-1

SECONDARY OUTCOMES:
Infarct growth between Day 7 and admission | At Day 7
  Infarct growth between Day 7 and admission on diffusion-weighted imaging
Early neurological deterioration | At Day 7
  Increment in NIHSS score by 2 points or more from admission
NIHSS score on Day 7 | At Day 7
  NIHSS score on Day 7
Good outcome | At 3 months
  mRS 0-2 at 3 months from stroke onset
mRS distribution at 3 months | At 3 months
  mRS distribution (assessed by shift analysis) at 3 months from onset
Ischemic stroke recurrence | At 3 months
  Ischemic stroke recurrence during 3 months from onset
Cost effectiveness of DAPT | Various (such as at 7 days or 3 months)
  Cost effectiveness analysis comparing DAPT to rt-PA

OTHER OUTCOMES:
Safety - symptomatic intracerebral hemorrhage | At 24 hours from the initial treatment
  symptomatic intracerebral hemorrhage
Safety - any intracranial bleeding | At 14 days from admission
  any intracranial bleeding
Safety - other hemorrhagic complications | At 14 days from admission
  other hemorrhagic complications
Safety - all-cause mortality | At 3 months
  all-cause mortality
Safety - cerebrovascular death | At 3 months
  cerebrovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Yuki Sakamoto, Principal Investigator — Nippon Medical School
Locations (27):
- Japan (27):
  - University of Yamanashi Hospital, Chūō
  - Fukuoka Red Cross Hospital, Fukuoka
  - Ota Memorial Hospital, Fukuyama
  - Kansai Medical University Hospital, Hirakata
  - Kagoshima City Hospital, Kagoshima
  - Kagoshima Medical Center, Kagoshima
  - Shioda Hospital, Katsuura
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - The Jikei University West Medical Center, Komae
  - Kawasaki Medical School Hospital, Kurashiki
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - The Jikei University Hospital, Minatoku
  - Kawasaki Medical School General Medical Center, Okayama
  - Kohnan Hospital, Sendai
  - Jichi Medical University Hospital, Shimotsuke
  - Nippon Medical School Tamanagayama hospital, Tama
  - Dokkyo Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Juntendo University Hospital, Tokyo
  - Nippon Medical School hospital, Tokyo
  - Science Tokyo Hospital, Tokyo
  - Tokyo Rosai Hospital, Tokyo
  - Tokyo Saiseikai Central Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Yamaguchi University Hospital, Ube
  - Juntendo University Urayasu Hospital, Urayasu

IPD SHARING:
Plan to Share IPD: Yes
On reasonable request.